CLINICAL TRIAL: NCT03906188
Title: Development and Validation of a Serious Game for Fibromyalgia Patients: Pre-experimental Study
Brief Title: Serious Game for Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Principal Investigator, ANA MARIA LARA PALMA, Principal Investigator, Universidad de Burgos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR 3/2018
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Fibromyalgia
Keywords: serious game; videogame
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LitEmotion group (Experimental): This group will play to LitEmotion video game.
  Interventions: Other: LitEmotion
- Control group (No Intervention): This group will no do receive any intervention with the video game

INTERVENTIONS:
Other: LitEmotion — LitEmotion is a serious video game programmed for helping managing emotions. The experimental group will play during 3 weeks while the control group will not play. The sample will play during 21 days, one session daily, around 45 minutes. After the 21 sessions the group will stop playing during 3 weeks. Therefore, the scales are done three times. In the very beginning (before playing), 21 days after playing, and, finally, 21 days no playing.
  Arms: LitEmotion group

SUMMARY:
Aim: To check the applicability of LitEmotion© in people with Fibromyalgia.

Design: randomized clinical trial, with pre, post and follow-up evaluation. Researchers and outcome evaluator blinded.

Method: The experimental group will play during three weeks to LitEmotion© videogame. The control group will not play.

DETAILED DESCRIPTION:
The study will be a longitudinal-transversal research work with two groups. Findings will us prove the correlation between a right management of emotions and the perception of pain, daily life activities and quality of sleeping.

Sample will be selected by following strict rules; people with no requirements will be dismissed.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosed
* Referred pain during the last month

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Health Assessment Questionnaire (HAQ) | Change from Baseline Independence Activities of the daily living up to 3 weeks
  The HAQ evaluates the performance in the activities of daily living.
Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline Independence Activities of the daily living up to 3 weeks
  The PSQI is an unreported measure which evaluate the quality of sleep.
Fibromyalgia Impact Questionnaire (FIQ) | Change from Baseline Independence Activities of the daily living up to 3 weeks
  The FIQ evaluates the quality of life in people with fibromyalgia.
Spanish Pain Questionnaire (SPQ). | Change from Baseline Independence Activities of the daily living up to 3 weeks
  The SPQ evaluates the kind of pain.

SECONDARY OUTCOMES:
Visual analogic scale (VAS) | Change from Baseline Independence Activities of the daily living up to 3 weeks
  The VAS evaluates the level of pain.
The spanish suggestibility inventory | Pre-assessment
  This inventory evaluates the level of suggestibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Burgos, Burgos, Spain

REFERENCES:
- [Background] Carmona, L. G., L.;Ballina, J.; Laffon, A. (2001). Proyecto EPISER 2000: prevalencia de las enfermedades reumáticas en la población española. Metodología, resultados del reclutamiento y características de la población. Revista Española de Reumatología, 28(1), 18-25.
- [Background] Esteve-Vives J, Rivera J, A Vallejo M; Grupo ICAF. [Assessment of functional capacity in fibromyalgia. Comparative analysis of construct validity of three functional scales]. Reumatol Clin. 2010 May-Jun;6(3):141-4. doi: 10.1016/j.reuma.2009.10.008. Epub 2010 Jan 27. Spanish. PMID 21794700
- [Background] Leavitt F, Katz RS, Golden HE, Glickman PB, Layfer LF. Comparison of pain properties in fibromyalgia patients and rheumatoid arthritis patients. Arthritis Rheum. 1986 Jun;29(6):775-81. doi: 10.1002/art.1780290611. PMID 3487324
- [Background] Rivera J, Gonzalez T. The Fibromyalgia Impact Questionnaire: a validated Spanish version to assess the health status in women with fibromyalgia. Clin Exp Rheumatol. 2004 Sep-Oct;22(5):554-60. PMID 15485007
- [Background] Rivera J, Alegre C, Ballina FJ, Carbonell J, Carmona L, Castel B, Collado A, Esteve JJ, Martinez FG, Tornero J, Vallejo MA, Vidal J. Documento de consenso de la Sociedad Espanola de Reumatologia sobre la fibromialgia. Reumatol Clin. 2006 Mar;2 Suppl 1:S55-66. doi: 10.1016/S1699-258X(06)73084-4. Epub 2008 Dec 10. No abstract available. Spanish. PMID 21794365